CLINICAL TRIAL: NCT01837511
Title: Analysis of the Incidence of Expression of Tumor Antigens MAGE-A3, MAGE-C2, NY-ESO-1, LAGE-1, WT1 and PRAME in Pathologically Proven Stage I, II and III Non-Small Cell Lung Cancer in Asiatic Patients
Brief Title: Analysis of the Incidence of Expression of Tumor Antigens in Pathologically Proven Stage I, II and III Non-Small Cell Lung Cancer(NSCLC) in Asiatic Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 109937
Record Dates: First submitted 2013-04-05; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Pathologically Proven Stage I, II and III Non-Small Cell Lung Cancer (NSCLC)
Keywords: Tumor antigens; Asiatic patients; Reverse Transciptase-Polymerase chain reaction (RT-PCR); Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cancer Group: Patients with pathologically proven stage I, II and III NSCLC.
  Interventions: Other: Data acquisition and analysis

INTERVENTIONS:
Other: Data acquisition and analysis — Tumor tissue samples submitted with a Patient and Tumor-Sample Characteristics. Form containing previously collected specific clinical data of patients with pathologically proven stage I, II and III NSCLC.

SUMMARY:
This study aims to investigate the expression of Melanoma-associated antigen 3 (MAGE-A3), Melanoma-associated antigen C2 (MAGE-C2), New York esophageal squamous cell carcinoma 1 (NY-ESO-1), L antigen family member 1 (LAGE-1), Wilms' tumor gene (WT1) and PRAME (PReferentially expressed Antigen of MElanoma) tumor antigens in a large number of pathologically proven stage I, II and III NSCLC samples of Asiatic patients.

DETAILED DESCRIPTION:
This study will be based upon the analysis of samples and patient-related data already available at the various investigation sites. There will be no study treatment and no study-specific procedure carried out on the patients.

Clinical data collected will include patient demographics (age, gender), Tumor, Node, Metastasis (staging system) [TNM stage], histopathologic description and the patient smoker status. Strict anonymity of patient data will be maintained.

This retrospective study is based upon the analysis of archived formalin-fixed paraffin-embedded tissue samples and patient-related data already available at the investigational site.

ELIGIBILITY:
Inclusion Criteria:

For inclusion of a tissue sample, all of the following criteria must be met:

* The patient had pathologically proven stage I, II or III NSCLC.
* All the data required are available from patient's records.
* Many patients may no longer be alive, or no longer be in contact with the investigation sites. Thus, patients will not be required to give their informed consent before inclusion in the study.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously collected samples and data of patients with pathologically proven stage I, II and III NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Determination of the expression of MAGE-A3, MAGE-C2, NY-ESO-1, LAGE-1, WT1 and PRAME antigens in tumor tissue from Asiatic patients with pathologically proven stage I, II or III NSCLC (as defined by the International Staging System). | Up to 6 months approximately.
Determination ofthe correlation of expression levels and co-expression patterns as detected by immunohistochemistry (IHC; protein expression) and as detected by RT-PCR (gene expression) for tumor antigens for which specific antibodies are available. | Up to 6 months approximately.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Singapore, Singapore
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul

REFERENCES:
- [Derived] Thongprasert S, Yang PC, Lee JS, Soo R, Gruselle O, Myo A, Louahed J, Lehmann FF, Brichard VG, Coche T. The prevalence of expression of MAGE-A3 and PRAME tumor antigens in East and South East Asian non-small cell lung cancer patients. Lung Cancer. 2016 Nov;101:137-144. doi: 10.1016/j.lungcan.2016.09.006. Epub 2016 Oct 5. PMID 27794402